CLINICAL TRIAL: NCT06354088
Title: Human Models of Selective Insulin Resistance: Alpelisib, Part I
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of California, Berkeley (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AAAU9636; K12DK133995 (NIH); K23DK140614 (NIH)
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Insulin Resistance; Prediabetic State; Overweight and Obesity; Non-Alcoholic Fatty Liver Disease
Keywords: Insulin resistance; Hyperinsulinemia; Non-Alcoholic Fatty Liver Disease; Hepatic steatosis; De novo lipogenesis; Glucose production
MeSH Terms: conditions — Insulin Resistance; Prediabetic State; Overweight; Obesity; Non-alcoholic Fatty Liver Disease; Hyperinsulinism; Fatty Liver | interventions — Alpelisib; Sodium Acetate; Glucose; delta inulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo then alpelisib (Insulin Sensitive group) (Experimental): On Study Visit 1, participants in the Insulin Sensitive (IS) group will undergo fasting and refed measurement of de novo lipogenesis (DNL) and endogenous glucose production (EGP) following a single dose of placebo. Then, 2-8 weeks later on Study Visit 2, participants will undergo measurement of DNL and EGP after a single dose of alpelisib 300 mg.
  Interventions: Drug: Alpelisib 300 mg; Drug: Placebo; Drug: [1-13C] sodium acetate; Drug: [6,6-2H2] D-glucose; Dietary Supplement: Nestlé BOOST Plus
- Alpelisib then placebo (Insulin Sensitive group) (Experimental): On Study Visit 1, participants in the Insulin Sensitive (IS) group will undergo fasting and refed measurement of de novo lipogenesis (DNL) and endogenous glucose production (EGP) following a single dose of alpelisib 300 mg. Then, 2-8 weeks later on Study Visit 2, participants will undergo measurement of DNL and EGP after a single dose of placebo.
  Interventions: Drug: Alpelisib 300 mg; Drug: Placebo; Drug: [1-13C] sodium acetate; Drug: [6,6-2H2] D-glucose; Dietary Supplement: Nestlé BOOST Plus
- Placebo then alpelisib (Insulin Resistant group) (Experimental): On Study Visit 1, participants in the Insulin Resistant (IR) group will undergo fasting and refed measurement of de novo lipogenesis (DNL) and endogenous glucose production (EGP) following a single dose of placebo. Then, 2-8 weeks later on Study Visit 2, participants will undergo measurement of DNL and EGP after a single dose of alpelisib 300 mg.
  Interventions: Drug: Alpelisib 300 mg; Drug: Placebo; Drug: [1-13C] sodium acetate; Drug: [6,6-2H2] D-glucose; Dietary Supplement: Nestlé BOOST Plus
- Alpelisib then placebo (Insulin Resistant group) (Experimental): On Study Visit 1, participants in the Insulin Resistant (IR) group will undergo fasting and refed measurement of de novo lipogenesis (DNL) and endogenous glucose production (EGP) following a single dose of alpelisib 300 mg. Then, 2-8 weeks later on Study Visit 2, participants will undergo measurement of DNL and EGP after a single dose of placebo.
  Interventions: Drug: Alpelisib 300 mg; Drug: Placebo; Drug: [1-13C] sodium acetate; Drug: [6,6-2H2] D-glucose; Dietary Supplement: Nestlé BOOST Plus

INTERVENTIONS:
Drug: Alpelisib 300 mg — All participants will ingest one dose of alpelisib 300 mg (2 x 150-mg overencapsulated tablets) on one of two study admissions.
  Other Names: Piqray
Drug: Placebo — All participants will ingest one dose of placebo (2 overencapuslated doses of microcrystalline cellulose) on one of two study admissions.
  Other Names: Placebo capsules
Drug: [1-13C] sodium acetate — All participants will receive continuous infusions of [1-13C] sodium acetate for up to 23 hours on both study visits in order to quantify de novo lipogenesis (DNL). (non-experimental)
  Other Names: C13A
Drug: [6,6-2H2] D-glucose — All participants will receive continuous infusions of [6,6-2H2] D-glucose for up to 15 hours on both study visits in order to quantify de novo lipogenesis (DNL). (non-experimental)
  Other Names: D2-glucose; D2G
Dietary Supplement: Nestlé BOOST Plus — All participants will ingest standardized mixed meals of Nestlé BOOST Plus on Study Day 1 and then smaller portions hourly x 8 hours on Study Day 2 of each study visit. (non-experimental)
  Other Names: Boost drink

SUMMARY:
The goal of this clinical trial is to understand how the blood sugar-lowering hormone insulin works in healthy adults versus those who are at risk for type 2 diabetes. The study will use a drug called alpelisib, which interferes with insulin's actions in the body, to answer the study's main question: does the liver continue to respond to insulin's stimulation of fat production even when it loses the ability to stop making glucose (sugar) in response to insulin. Researchers will compare the impact of single doses of both alpelisib and placebo (inert non-drug) in random order (like flipping a coin) in study participants. Participants will be asked to stay twice overnight in the hospital, take single doses of alpelisib and placebo (one or the other on each of the two hospital stays), and receive intravenous (into the vein) infusions of non-radioactive "tracer" molecules that allow researchers to measure the production of glucose (sugar) and fats by the liver. Measurements will be done both overnight, while participants are asleep and fasting (not eating or drinking other than water) and while consuming a standardized diet of nutritional beverages during the following day.

The objective is to evaluate the effect of lowering insulin levels, while maintaining constant mild hyperglycemia, on plasma glucose and lipid levels.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is an under-appreciated complication of lipid dysmetabolism in type 2 diabetes (T2DM). Although it appears that insulin resistance (IR) is a mechanism common to both, the mechanisms linking IR to unhealthy fat accumulation in liver remains unclear. "Pure" IR would be expected to disinhibit hepatic glucose production while dampening hepatic triglyceride (TG) biosynthesis, but the excessive hepatic de novo lipogenesis (DNL) of IR-associated MASLD suggests that hepatic IR is "selective." However, the concept of IR selectivity is controversial, and because of clinical heterogeneity, lead-time discrepancies, co-morbidities, and medication effects, parsing out this pathophysiologic conundrum in humans is challenging. The investigators plan to test whether the multifactorial IR in patients at risk of T2DM/MASLD is selective by determining if inducing a discrete, "pure" form of IR, via pharmacologic inhibition of phosphoinositide-3-kinase (PI3K) with alpelisib, versus placebo, attenuates excessive DNL. Investigators will also study this question in healthy, insulin-sensitive (IS) volunteers.

Participants in this randomized crossover trial will be admitted twice to the inpatient clinical research unit. During each admission, they will take a dose of either alpelisib or placebo (in randomized order) in the evening and receive infusions of [13C] sodium acetate and [2H] D-glucose to measure DNL and endogenous glucose production (EGP), respectively, during an overnight fast. DNL measurement will then continue during the following day during 8 hours of standardized mixed-meal feedings. Blood will be drawn at defined intervals for determining levels of glucose, insulin, lipids including triglycerides and free fatty acids, and tracer/tracee enrichments for the stable-isotope tracers. There will be a 2-8-week hiatus for drug washout between the two inpatient study admissions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-70 years, using highly effective contraception if of childbearing potential
2. Able to understand written and spoken English and/or Spanish
3. Body mass index of:

   * For Group IS: BMI 18-25 kg/m2
   * For Group IR: BMI 30-45 kg/m2
4. Evidence of insulin sensitivity or insulin resistance:

   * Insulin sensitive (for Group IS) defined as all of the following: (1) Fasting serum insulin ≤ 10 µIU/mL, (2) Absence of dysglycemia (fasting plasma glucose < 100 mg/dL and hemoglobin A1c < 5.7%), (3) Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) score < 2.5, and (4) Fibrosis-4 (FIB-4) score < 1.3
   * Insulin resistant (for Group IR) defined as fasting serum insulin ≥ 13 µIU/mL plus at least one of the following: (1) Presence of prediabetic state (fasting plasma glucose 100-125 mg/dL and/or hemoglobin A1c 5.7-6.4%), and/or HOMA-IR ≥ 2.5

Exclusion Criteria:

1. Inability to provide informed consent in English or Spanish
2. Concerns arising at screening visit:

   * Abnormal vital signs: (1) Systolic blood pressure < 90 mm Hg or > 160 mm Hg and/or (2) Diastolic blood pressure < 55 mm Hg or > 100 mm Hg and/or (3) Abnormal resting heart rate < 55 bpm (except at PI's discretion) or ≥ 110 bpm
   * Abnormal screening serum electrolytes judged by the PI to be potentially clinically significant, including liver function abnormalities (either of the following): (1) Transaminases (AST or ALT) > 3.0 x the upper limit of normal and/or (2) Total bilirubin > 1.25 x the upper limit of normal
   * Laboratory evidence of diabetes mellitus: (1) Hemoglobin A1c ≥ 6.5%, and/or (2) Fasting plasma glucose ≥ 126 mg/dL
3. Reproductive concerns i. Positive qualitative β-hCG (i.e., pregnancy test) in women of childbearing potential ii. Women currently pregnant iii. Women currently breastfeeding
4. Concerns related to glucose metabolism

   * History of having met any of the American Diabetes Association's definitions of diabetes mellitus (i.e., overt diabetes)
   * History of gestational diabetes mellitus within the previous 5 years
   * Use of most antidiabetic medications (other than metformin) within the 90 days prior to screening: thiazolidinediones, sulfonylureas, meglitinides, dipeptidyl peptidase-4 (DPP4) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists, sodium-glucose cotransporter-2 (SGLT2) inhibitors, amylin mimetics, acarbose, insulin iv. Clinical concern for absolute insulin deficiency (e.g., type 1 diabetes, pancreatic disease)
5. Concerns related to lipid metabolism

   * Known diagnoses of familial hypercholesterolemia, familial combined hyperlipidemia, or familial hyperchylomicronemia in the participant or a first-degree relative
   * Use of certain lipid-lowering drugs within 14 d prior to screening visit: fibrates (e.g., fenofibrate, gemfibrozil), prescription-strength omega-3 fatty acids (e.g., icosapent ethyl), high-dose niacin (>100 mg daily)
6. Known, documented history, at the time of screening, of any of the following medical conditions:

   * Significant cardiovascular diseases (N.B. uncomplicated hypertension is not exclusionary)
   * Severe liver disease, including advanced fibrosis (e.g., fibrosis score F3-F4 by vibration-controlled transient elastography) and cirrhosis
   * Psychiatric diseases causing functional impairment that: (1) Are or have been decompensated within 1 year of screening, and/or (2) Require use of anti-dopaminergic antipsychotic drugs associated with significant weight gain/metabolic dysfunction (e.g., clozapine, olanzapine)
   * Venous thromboembolic disease (deep vein thrombosis or pulmonary embolism) or any required use of therapeutic anticoagulation
   * Bleeding disorders, including due to anticoagulation, or significant anemia (see above)
   * Active malignancy, or hormonally active benign neoplasm, except allowances for non-melanoma skin cancer and differentiated thyroid cancer (Stage I only)
7. Clinical concern for increased risk of volume overload, including due to medications and/or heart/liver/kidney problems, as listed above
8. Use of oral or parenteral corticosteroids (at greater than prednisone 5 mg daily, or equivalent) for more than 3 days within the previous 30 days; topical and inhaled formulations are permitted
9. History of certain weight-loss (bariatric) surgery, including:

   * Roux-en-Y gastric bypass
   * Biliopancreatic diversion
   * Restrictive procedures (lap band, sleeve gastrectomy) performed within the past 6 months
10. Clinical concern for alcohol overuse based on chart review and/or by recruit's report of more than 14 standard drinks per week for males or more than 7 standard drinks per week for females
11. Regular use of tobacco, either daily or an average of at least 1 cigarette per day, and/or nicotine vaping more than 1 day per week
12. Clinical concern for use of illicit drugs other than marijuana or lawfully prescribed medications based on recruit's report, chart review, and point-of-care urine drug test at screening
13. History of or ongoing febrile illness within 30 days of screening
14. Any other disease or condition or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
15. Known allergy/hypersensitivity to any component of the medicinal product formulations (including soy, cow dairy, or gluten), other biologics, venipuncture materials, plastics, adhesive or silicone, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
16. Dietary restrictions (e.g., vegan, kosher, halal) on gelatin present in overencapsulation
17. Concurrent enrollment in another clinical study of any investigational drug/biologic therapy within 6 months prior to screening or within 5 half-lives of an investigational agent or biologic, whichever is longer.

    * Prior participation in other studies led by Dr. Cook (PI) is excluded from this prohibition according to his medical/scientific judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hepatic de novo lipogenesis (DNL) (absolute value) | Up to 24 hours after dosing
  Percent incorporation of newly synthesized fatty acids into plasma or VLDL TG. During both inpatient (overnight) study visits, starting after investigational agent dose.
  units: %
Hepatic de novo lipogenesis (DNL) (relative value) | Up to 24 hours after dosing
  Percent incorporation of newly synthesized fatty acids into plasma or VLDL TG. During both inpatient (overnight) study visits, starting after investigational agent dose.
  unit: fold difference and/or ∆% versus other group
Endogenous glucose production (EGP) (absolute value) | Up to 15 hours after dosing
  Calculated from D2G tracer enrichment by the Steele equations. During both inpatient (overnight) study visits, starting after investigational agent dose.
  units: mg/kg/min
Endogenous glucose production (EGP) (relative value) | Up to 15 hours after dosing
  Calculated from D2G tracer enrichment by the Steele equations. During both inpatient (overnight) study visits, starting after investigational agent dose.
  units: fold difference and/or ∆% versus other group

SECONDARY OUTCOMES:
Serum insulin level | Approximately 11-19 hours after dosing
  Serum insulin levels in response to placebo vs alpelisib following an overnight fast and then hourly during refeeding.
  During Study Day 2 of both study visits, starting after investigational agent dose.
  units: µIU/mL
Plasma glucose level | Approximately 11-19 hours after dosing
  Plasma glucose levels in response to placebo vs alpelisib following an overnight fast and then hourly during refeeding.
  During Study Day 2 of both study visits, starting after investigational agent dose.
  units: mg/dL
Triglycerides level | Approximately 11-19 hours after dosing
  (Serum or plasma) triglyceride levels in response to placebo vs alpelisib following an overnight fast and then hourly during refeeding.
  During Study Day 2 of both study visits, starting after investigational agent dose.
  units: mg/dL
Free fatty acids level | Approximately 11-19 hours after dosing
  (Serum or plasma) triglyceride levels in response to placebo vs alpelisib following an overnight fast and then periodically during refeeding.
  During Study Day 2 of both study visits, starting after investigational agent dose.
  units: mmol/L
Glucose kinetics: rate of appearance (absolute value) | Up to 15 hours after dosing
  Calculated from D2G tracer enrichment by the Steele equations. During both inpatient (overnight) study visits, starting after investigational agent dose.
  units: mg/kg/min
Glucose kinetics: rate of appearance (relative value) | Up to 15 hours after dosing
  Calculated from D2G tracer enrichment by the Steele equations. During both inpatient (overnight) study visits, starting after investigational agent dose.
  units: fold difference and/or ∆% versus other group
Glucose kinetics: rate of disappearance (absolute value) | Up to 15 hours after dosing
  Calculated from D2G tracer enrichment by the Steele equations. During both inpatient (overnight) study visits, starting after investigational agent dose.
  units: mg/kg/min
Glucose kinetics: rate of disappearance (relative value) | Up to 15 hours after dosing
  Calculated from D2G tracer enrichment by the Steele equations. During both inpatient (overnight) study visits, starting after investigational agent dose.
  units: fold difference and/or ∆% versus other group

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes